CLINICAL TRIAL: NCT06904989
Title: Implementation and Evaluation of a New Cancer Rehabilitation Process for the Assessment and Treatment of Chemotherapy-Induced Foot Neuropathy - A Collaborative Project Between Oncology Clinic and Orthopedic Technology Department 2.0.
Brief Title: A New Cancer Rehabilitation Process for Chemotherapy-Induced Foot Neuropathy Using Orthopedic Devices
Acronym: FOTNEV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-05490-01
Record Dates: First submitted 2025-03-10; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-11

CONDITIONS: Polyneuropathy; Breast Cancer
Keywords: Chemotherapy-Induced Peripheral Neuropathy (CIPN); Oncology Rehabilitation; Orthopedic Intervention; Breast Cancer; Orthopedic Insoles
MeSH Terms: conditions — Polyneuropathies; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard orthopedic treatment (Active Comparator): Patients provided with customized shoes and insoles for outdoor use
  Interventions: Device: Standard Treatment
- Silicone orthose (Experimental): Patients provided with customized shoes and insoles for outdoor use + a specialized sock for indoor use.
  Interventions: Device: Silicone orthosis

INTERVENTIONS:
Device: Silicone orthosis — in addition to standard treatment, shoe and insole treatment, a new type of treatment for CIPN is being evaluated, a silicone orthosis.The silicone orthosis consists of a half-sock designed for indoor use.
  The participants feet are examined, and the foot shape is scanned barefoot using a three-dimensional foot scanner from Volumental. This is performed to use a basis for manufacturing individual silicone orthoses. Activity measurement with an activity sensor, attached to the thigh with tape, is planned for two weeks after receiving the assistive device.
  Participants who receive a silicone orthosis are asked to keep a diary of how much they have used it. The follow-up takes place at the Oncology Department 3-6 weeks after the participant has received the assistive device.
  Arms: Silicone orthose
Device: Standard Treatment — The standard treatment is that patients are provided with customized insoles and shoes. Foot status is recorded during the orthopedic technical assessment at OTA, identifying signs of neuropathy, impaired blood circulation, foot deformities, and skin pathologies. A modified version of the validated D-Foot instrument is used to assess the risk of foot ulcers, especially in diabetic patients. The evaluation also includes lower extremity function, gait abnormalities, and existing footwear and insoles.
  Differences in foot anthropometry are compared between scanned foot measurements of the study group and those of a control group representing a female Swedish normal population.
  ActivePal is a reliable method for measuring and classifying activity levels. Activity measurement is conducted over two weeks.
  Arms: Standard orthopedic treatment

SUMMARY:
The goal of this clinical study is to evaluate a new process for assessing and alleviating chemotherapy-induced peripheral neuropathy in the feet in patients treated with chemotherapy for early stage breast cancer. It will also compare two orthopedic interventions for symptom relief. The main questions it aims to answer are:

Can an orthopedic silicone orthosis reduce chemotherapy-induced peripheral neuropathy symptoms in the feet? How does the effectiveness of the silicone orthosis compare to standard orthopedic treatment with insoles and shoes?

Participants will:

Use either a silicone orthosis or standard orthopedic treatment Have contact with the clinic for assessments and follow-ups Report their symptoms and functional improvements over time

DETAILED DESCRIPTION:
Background and Rationale

This study aims to develop and evaluate a structured multidisciplinary rehabilitation process for assessing and managing chemotherapy-induced peripheral neuropathy in the feet. The project establishes a new collaboration between the Oncology Department and the Department of Orthopedic Technology at Sahlgrenska University Hospital, integrating an orthopedic approach into cancer rehabilitation.

Chemotherapy-induced peripheral neuropathy is a common side effect of chemotherapy, affecting 50-90% of patients undergoing cancer treatment. Symptoms such as numbness, tingling, pain, and sensory loss in the feet can lead to chronic discomfort, impaired balance, and reduced quality of life. Despite its prevalence, there are no standardized guidelines for grading or managing chemotherapy-induced peripheral neuropathy within rehabilitation. Additionally, structured follow-up for chemotherapy-induced peripheral neuropathy after chemotherapy is lacking in Sweden, and there are limited effective treatment options available.

This research project aims to develop a structured process for assessing and managing chemotherapy-induced peripheral neuropathy in the feet and to evaluate two orthopedic interventions:

* Current standard treatment - customized insoles and orthopedic shoes.
* A novel intervention - a silicone orthosis, designed as a soft, sock-like device for indoor use.

Although silicone orthoses have been introduced in limited clinical settings in Sweden, their effectiveness for chemotherapy-induced peripheral neuropathy remains untested. This study seeks to evaluate whether this new intervention can alleviate symptoms and improve mobility and quality of life for breast cancer patients experiencing chemotherapy-induced peripheral neuropathy .

Study Objectives

The overall aim is to establish and evaluate a new process for assessing and alleviating symptoms in the feet through orthopedic technology. Specifically, the study will:

* Compare the effectiveness of two orthopedic interventions (custom insoles vs. silicone orthosis).
* Investigate patient-reported outcomes regarding symptom relief, quality of life, and functional mobility.

Study Design and Methodology The study consists of a pilot phase with, followed by a potential randomized controlled trial if preliminary results are promising. This pilot study will include 40 participants, divided equally between the two intervention groups. It is conducted at Sahlgrenska University Hospital, involving a multidisciplinary collaboration between the Oncology Department and the Orthopedic Technology Department .

Step 1: Diagnosis and Assessment Patients with chemotherapy-induced peripheral neuropathy in the lower extremities (feet) following breast cancer treatment will be assessed using a standardized grading system based on the Common Terminology Criteria for Adverse Events as well as a symptom questionnaire. Patients will also complete self-reported quality-of-life assessments as well as the EQ-5D scale and undergo 3D foot scanning to measure foot morphology and structural differences compared to the general population. Medical records will be reviewed to collect demographic and clinical variables (age, cancer status, chemotherapy regimen, comorbidities, smoking status, Body Mass Index).

Step 2: Orthopedic Interventions

Patients will be randomly assigned to one of two intervention groups:

Group 1: Receives customized orthopedic insoles and shoes, the current standard treatment for diabetic neuropathy.

Group 2: Receives a silicone orthosis, a novel sock-like support designed for indoor use.

All participants will receive guidance on footwear selection and be provided with seamless socks to minimize pressure on sensitive areas.

All patients will also be examined with

* D-Foot: A validated and reliable instrument for structured foot examination, primarily used in diabetic foot assessments.
* 3D foot scanning (Volumental scanner): Provides highly accurate foot measurements with a ±1 mm error margin.

Step 3: Activity Monitoring

To objectively assess mobility and functional changes, patients will wear an activity tracker (Active Pal) attached to their leg using skin-friendly tape for two weeks. The device records data on:

* Time spent sitting, standing, walking, or lying down.
* Step count and movement patterns. Patients in the silicone orthosis group will also maintain a daily usage diary to document how often they wear the device.

Step 4: Follow-Up and Outcome Evaluation

Follow-up assessments will occur 3-6 weeks post-intervention, conducted by oncology nurse or doctor via:

* Repeat symptom grading (CTCAE).
* Self-reported questionnaires on foot health and quality of life.
* Semistructured interviews evaluating patients' experiences with their assigned intervention.

Interviews will explore:

* Perceived symptom relief and comfort.
* Impact on daily activities and mobility.
* Satisfaction with the provided intervention.
* The follow-up can be conducted in person, via phone, or digitally and is estimated to take approximately 45 minutes.

Scientific Questions

The study aims to answer the following key research questions:

* What is the prevalence and severity of chemotherapy-induced peripheral neuropathy in the feet among the patients?
* How does chemotherapy-induced peripheral neuropathy affect self-reported quality of life (EQ-5D scores)?
* What is the foot status (e.g., structural and functional characteristics) in affected patients?
* Are there foot morphology differences between chemotherapy-induced peripheral neuropathy patients and the general female population?
* Does the type of orthopedic aid influence activity levels and mobility?
* How does chemotherapy-induced peripheral neuropathy impact patients' daily lives?
* Are there differences in patient experience and perceived effectiveness between the two orthopedic interventions?

Expected Impact

If successful, this study will:

* Provide new insights into the effectiveness of orthopedic aids for chemotherapy-induced peripheral neuropathy -related foot symptoms.
* Establish a structured assessment process for chemotherapy-induced peripheral neuropathy in oncology rehabilitation.
* Improve patient quality of life by offering evidence-based interventions for symptom relief.
* Lay the groundwork for a larger randomized controlled trial to confirm findings and influence future clinical guidelines.

By bridging the gap between oncology and orthopedic technology, this project aims to enhance rehabilitation strategies for cancer survivors dealing with long-term neuropathic complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer receiving treatment at the Oncology Department, Sahlgrenska University Hospital (SU).
* Have undergone treatment with taxanes.
* Aged 18 years or older.
* Able to understand spoken and written Swedish.
* Patients who can ambulate with or without assistive walking devices.
* CTCAE grading above 2 at a medical visit after completing treatment.

Exclusion Criteria:

* Bilateral amputation at the thigh level.
* Previously diagnosed neurological disease or neurological impairment affecting the feet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Change in foot neuropathy grade after 3-6 weeks of using the silicone orthosis. | At baseline and after three to six weeks after treatment initiation
  Neuropathy severity will be assessed using the NCI-CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) version 5.0, a standardized tool for grading adverse events related to cancer treatment, including chemotherapy-induced peripheral neuropathy (CIPN).
  CIPN is classified into five grades based on motor, sensory, and autonomic symptoms:
  Grade 1 (Mild): Asymptomatic or mild symptoms with no significant impact on daily activities.
  Grade 2 (Moderate): Symptoms affecting daily activities but not requiring intervention.
  Grade 3 (Severe): Symptoms severely limiting self-care and daily functions. Grade 4 (Life-threatening): Disabling symptoms requiring urgent intervention. Grade 5 (Fatal): Death related to adverse effects. Higher grades indicate more severe neuropathy and are used to monitor patient safety, adjust treatments, and evaluate drug toxicity in clinical oncology settings.
Change in Change in physical activity level after 3-6 weeks of using the silicone orthosis. | During two weeks after initiation of treatment
  The device records movement patterns and classifies activity into three main categories:
  Sedentary time (e.g., sitting or lying down) Standing time Stepping time (walking or other movement) The data is collected over a period of two weeks, allowing researchers to analyze changes in mobility and activity levels. The first few days serve as an adaptation phase, after which the measurements are expected to reflect habitual daily activity. The digital activity data is often combined with patient diaries to provide a more comprehensive analysis of movement patterns and intervention effects.
Change in foot neuropathy symptoms after 3-6 weeks of using the silicone orthosis. | At baseline and after 3-6 weeks after initiation of treatment.
  The modified CIPN20 questionnaire is a tool for assessing chemotherapy-induced peripheral neuropathy symptoms and their impact on daily life. It consists of 20 items, covering sensory (9 items), motor (8 items), and autonomic (3 items) domains.
  Each item is rated on a 5-point Likert scale:
  0 = Not at all
  1. = A little
  2. = Somewhat
  3. = Quite a bit
  4. = Very much Higher scores indicate more severe symptoms and functional impairment. The scores can be analyzed separately for each domain or as a total CIPN burden, making the questionnaire useful for monitoring symptom progression and evaluating treatment effects.

SECONDARY OUTCOMES:
Change in self reported quality of life in patients with foot neuropathy after 3-6 weeks of using the silicone orthosis. | At enrollment and after three to six weeks after treatment initiation
  The EQ-5D is a standardized tool for measuring health-related quality of life (HRQoL). It provides a simple, generic measure of health status and is used in both clinical and research settings to assess treatment outcomes and patient well-being.
  Structure and Scoring The EQ-5D consists of five dimensions, each rated on a 5-point scale: Mobility (ability to walk) Self-care (ability to wash/dress oneself) Usual activities (work, study, household tasks, etc.) Pain/discomfort Anxiety/depression Each dimension is scored from 1 (no problems) to 5 (extreme problems), generating a unique health profile that can be converted into a single index score using country-specific value sets. Additionally, EQ-5D includes a Visual Analog Scale (VAS), where patients rate their overall health from 0 (worst imaginable health) to 100 (best imaginable health).
  The EQ-5D is useful for tracking changes in health status over time, comparing treatment effects, and informing health economic ev
Comparisons of foot status based on a structured foot examination. | The comparison is based on a one-time examination at enrollment.
  Foot status is recorded during the orthopedic technical assessment. The examination identifies signs of neuropathy, impaired blood circulation, foot deformities, skin pathologies, and a history of ulcers or amputations using a modified version of D-Foot. D-Foot is a validated and reliable instrument for structured foot examinations, primarily used to identify diabetic patients at increased risk of foot ulcers. In addition to foot status, lower extremity function, gait abnormalities, and existing footwear and insoles are documented
Differences in foot anthropometry between study group and a control group representing a female Swedish normal population | The comparison is based on a one-time examination at enrollment.
  Differences in foot anthropometry are compared between scanned foot measurements of the study group and those of a control group representing a female Swedish normal population. Based on 3D foot scanning of the participant's feet, measurements such as foot length, foot width, and toe height are obtained. The Volumental scanner has a measurement error margin of 1 mm.

OTHER OUTCOMES:
Patients' experiences using orthotic devices in order to relieve symptoms of CIPN in the feet after treatment for early-stage breast cancer. | A one-time occasion 6-10 weeks after enrollment.
  Semi-structured interviews are planned. Focusing on the experience of using an orthotic device that intends to relieve CIPN-symptoms. An interview guide has been developed based on prior research and clinical experience. Each interview is scheduled to last 30-45 minutes. Interviews will be recorded, transcribed and numbered.
Patients' experiences of living with CIPN after treatment for early-stage breast cancer | A single assessment conducted before the start of treatment
  Results are expected to answer how CIPN is experienced and affects various aspects of daily life, both individually and collectively. What is the discomfort in daily life, and are any self-care strategies used to alleviate symptoms? Semi-structured interviews are planned, focusing on the experience of living with CIPN in the feet. An interview guide has been developed based on prior research and clinical experience. Each interview is scheduled to last 30-45 minutes. Interviews will be recorded, transcribed and numbered.

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Hellstrand Tang, Orthopedic engineer, Principal Investigator — Vastragotaland regionen
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No